CLINICAL TRIAL: NCT00771056
Title: Phase II Study to Evaluate the Tolerability and Efficacy of Treatment of Previously Untreated B-Cell Chronic Lymphocytic Leukemia (B-CLL) Patients With Hydroxychloroquine.
Brief Title: Hydroxychloroquine in Untreated B-CLL Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study suspended while data is reviewed for safety and efficacy.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Kanti Rai, MD, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-088
Record Dates: First submitted 2008-10-08; First posted 2008-10-10 (Estimated); Results first posted 2016-07-26 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
Keywords: untreated
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydroxychloroquine (Experimental): Hydroxychloroquine 400 mg po daily for up to one year.
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — 400mg by mouth daily x 1 year
  Other Names: Plaquenil

SUMMARY:
Eligible CLL patients who sign an informed consent will be started on hydroxychloroquine 400mg po daily for up to one year. They will be monitored for disease status as well as adverse reactions after two weeks and then every 4 weeks. Ophthalmologic exams is required at baseline and every 6 months or sooner if the patient develops any visual disturbances.

DETAILED DESCRIPTION:
This is a single-center, open-label, single arm Phase 2 study evaluating the feasibility, and efficacy of treating CLL subjects with hydroxychloroquine. The study schema and schedule of events are as follows:

Prior to beginning hydroxychloroquine:

* Blood samples to be taken.
* Baseline tests confirming diagnosis of CLL as defined above (if not already obtained in records)
* Physical exam performed
* Either six months prior or 4 weeks within starting HCQ ophthalmologic exam documented
* Days 1-365 subject takes hydroxychloroquine 400mg/day
* At 2 weeks: CBC and chemistry
* Every 4 weeks: CBC, chemistry, history (including the inquiry about the presence or absence of visual symptoms) and physical exam.
* Starting at 4 weeks: blood samples taken for laboratory companion studies taken at office visit every 8 weeks.
* At 6 months (+ or - 30 days): subject will have follow up ophthalmologic exam). This will also be done in the presence of any visual/ocular symptoms.

All subjects must meet the selection criteria for registration in this study. All subjects must have a peripheral blood sample submitted. It is estimated that approximately 70 subjects will be screened. The anticipated accrual period is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Flow cytometry confirmed B-CLL
* No prior chemotherapy or immunotherapy
* Performance status 0-2
* Age > 18 years old
* If childbearing age, woman you must be willing to use birth control for length of hydroxychloroquine use
* Must have capacity to consent for study and sign consent form
* Asymptomatic CLL not requiring treatment at time of study entry

Exclusion Criteria:

* Pregnancy
* Significant optic nerve pathology as documented by an opthalmologic exam
* Hypersensitivity to 4-aminoquinoline compound
* Patients taking cardiac glycosides and cyclosporine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanti R Rai, MD, Principal Investigator — NSLIJ
Locations (1):
- Long Island Jewish Medical Center CLL Research and Treatment Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to contact each individual patient (participant in the trial) and inform hem/her of results of this trial as it affects each one of them.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from April 2009 through termination December 2011. Patients were identified and enrolled in the CLL Research and Treatment Program where they already were being seen for care of their CLL.
Period: Overall Study
Arm/Group | Hydroxychloroquine
Started | 23
Completed | 18
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Hydroxychloroquine
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 59 [44 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response
Description: Percentage of participants with a reduction of the absolute lymphocytic count- ALC
Time Frame: 1 yr
Measure: Number; unit: percentage of participants
Arm/Group | Hydroxychloroquine
Number analyzed (Participants) | 23
percentage of participants | 54.4

2. Secondary Outcome: Time to Next Treatment
Description: number of months to time from last HCQ dose to next CLL treatment
Time Frame: 1 yr
Population: only analyzed for participants that were treated within one year post last dose of hydroxychloroquine dose
Measure: Mean (Full Range); unit: months
Arm/Group | Hydroxychloroquine
Number analyzed (Participants) | 3
months | 4.3 [2 to 7]

ADVERSE EVENTS:
Time Frame: Adverse event reporting wil be reported if applicable as subjects are monitored on a monthly basis.
Description: Subjects were monitored monthly by physician for adverse events from hydroxychloroquine.
Arm/Group | Hydroxychloroquine
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes